CLINICAL TRIAL: NCT01359839
Title: Relaxation-Response Based Cognitive Behavioral Therapy Group for Depressed Chinese Patients in the Community
Brief Title: Effectiveness of a Relaxation-Response Based Cognitive Behavioral Therapy Group for Depressed Chinese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Albert Yeung, Psychiatrist, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2009P002557
Record Dates: First submitted 2011-05-23; First posted 2011-05-25 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Relaxation Response Mind Body Intervention (Experimental): The Relaxation Response (RR) Mind Body Intervention Arm receives the Behavioral: Relaxation Response and Cognitive Behavioral Therapy Intervention which is a RR based Mind Body Group consisting of 1½ hour group classes held weekly for 8 weeks, in a conference room at the health center.
  Interventions: Behavioral: Relaxation Response and Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Relaxation Response and Cognitive Behavioral Therapy — This is a group format which will meet once per week and teach the techniques of cognitive behavioral therapy as well as relaxation response meditation.

SUMMARY:
The goal of this research is to evaluate whether group therapy combining Relaxation Response (RR) training and Cognitive Behavioral Therapy (CBT) in a group format merits further investigation in the treatment of Major Depressive Disorder (MDD). Specifically, the primary aim of this waitlist-controlled study is to gather preliminary data evaluating the effectiveness of RR-CBT group as treatment for patients with current MDD or a history of MDD, including patients who continue to be depressed despite taking antidepressants and patients who choose not to take antidepressants due to the fear of side effects and/or for personal reasons.

DETAILED DESCRIPTION:
The Epidemiological Catchment Area Study found that the lifetime prevalence of depression ranged from 5-8%. A more recent assessment found that the lifetime prevalence of Major Depression is greater than previously estimated, with 12% of men and 21% of women suffering from the disorder. The point prevalence for major depression (MDD) is approximately 13% for women and 8% for men.

Despite the growing number of marketed antidepressants, between 19-34% of depressed patients still do not respond to acute antidepressant treatment, 29-46% may fail to achieve and sustain a full remission, and between 15-50% will have a recurrence of depression despite continuous antidepressant treatment. The side effects of antidepressants are common and account significantly for premature treatment discontinuation.

When a first line treatment for depression fails, clinicians often choose to increase the dosage, or augment with a second agent, prior to considering switching agents altogether. Combination of an SSRI/SNRI with other agents such as tricyclic antidepressants (TCAs) or lithium are examples of popular strategies. In many instances, augmentation with multiple psychotropic agents may not be desirable, because of risk of side effects or drug-drug interactions.

In view of their benign adverse effect profiles, non-pharmacological interventions such as psychotherapy and mind-body intervention have been used to augment treatment for treatment resistant depressed patients. Preliminary studies have shown that meditation is beneficial for the treatment of depression.

Research has shown that Cognitive Behavioral Therapy(CBT) is effective for both acute and maintenance psychotherapies. In addition, CBT has been shown not only to induce acute remission, but to provide prophylaxis against relapse and recurrence. CBT may impart skills that patients can continue to use after acute treatment ends.

This is a pilot study to investigate the effectiveness of group therapy combining Relaxation Response (RR) training and CBT for depressed Chinese in the community.

ELIGIBILITY:
Inclusion criteria

* Men and women between the ages of 18 and 65 years;
* Chinese Americans
* Satisfy DSM-IV criteria for current Major Depressive Disorder (MDD), or have a history of MDD, prior to the initiation of RR-CBT group treatment, as determined by the SCID interview;
* HAM-D-17 baseline score ≥14; and
* Have not had CBT treatment and have not started other forms of mind/body intervention in the past 3 months.

Exclusion criteria

* Patients with primary diagnosis other than MDD and/or do not have a history of MDD;
* Any history of psychosis, mania, or severe cluster B personality disorder;
* Conditions that may make it difficult to conclusively determine that depressive symptoms are the result of MDD or having a history of MDD and not some other condition, including any form of substance abuse or dependence within the last 6 months, relevant medical conditions that may be the medical basis of a depression including epilepsy, history of an abnormal EEG, severe head trauma, or stroke;
* Medical conditions that would preclude entry into a clinical trial, including serious uncontrolled medical conditions (e.g. poorly controlled diabetes, severe congestive heart failure), or other medical conditions that have not been stable for a minimum of 3 months;
* Confounding treatments, such as current ongoing treatment other than what is provided by South Cove for depression; plans to receive confounding treatments (including the treatment of endocrinopathies); or starting new mind-body interventions including Qigong, mindfulness training, muscle relaxation training, etc.;
* Electroconvulsive therapy (ECT) during the last year; and
* Current active suicidal or self-injurious potential necessitating immediate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Improvement in depressive symptoms | Eight Weeks
  Improvement in depressive symptoms will be assessed using the resulting scores from the questionnaire forms Q-LES-Q-SF (Quality of Life Enjoyment Satisfaction Questionnaire Short Form) and the HAM-D (Hamilton Depressive Scale).

SECONDARY OUTCOMES:
Score on the Q-LES-Q-SF | Eight Weeks
  Quality of Life Enjoyment Satisfaction Questionnaire Short Form

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, Principal Investigator — Massachusetts General Hospital; Herbert Benson, MD, Study Director — Massachusetts General Hospital; John Denninger, MD, PhD, Study Director — Massachusetts General Hospital; Gregory Fricchione, MD, Study Director — Massachusetts General Hospital
Locations (1):
- South Cove Community Health Center, Boston, Massachusetts, United States